CLINICAL TRIAL: NCT01425957
Title: Identification of Biomarkers Sensitive to Disease Progression in Patients With Mild Cognitive Impairment: a Two-part Clinical Study. PartA: Multisite MRI Acquisition, Protocol Harmonization. PartB: Identification of Biomarkers Sensitive to Disease Progression in Patients With Mild Cognitive Impairment: a Clinical Study
Brief Title: Identification of Biomarkers Sensitive to Disease Progression in Patients With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qualissima (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WP5P001; 2011-A00985-36 (Other: ID-RCB from AFSSAPS)
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: MILD COGNITIVE IMPAIRMENT
Keywords: MEMORY and COGNITIVE IMPAIRMENT; ALZHEIMER DISEASE CONVERSION; Amyloid beta-Peptides
MeSH Terms: conditions — Cognitive Dysfunction; Plaque, Amyloid | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCI Patient with Lumbar puncture (Other): PartB: Patients affected by amnestic Mild Cognitive Impairment (aMCI).
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — All the patients will be divided in two groups based on their Aβ 1-42 levels measured in the cerebro-spinal fluid obtained form a lumbar puncture: in low Aβ1-42 (positive aMCI patients CSFP) and high Aβ1-42 (Negative aMCI patients CSFN). The threshold of Aβ1-42 used to divide the patient will be 500 (ng/L) based on Sjogren criteria (2001).
  Timeframe of lumbar punctures: every 18 months during 2 years (T0 and T18) or 3 years (T0, T18 and T36).
  Other Names: Cerebrospinal fluid puncture

SUMMARY:
THE STUDY WILL BE A TWO-PART RESEARCH

PART A and PART A extended:

1. To implement a "common" MRI acquisition protocol in multiple centers across Europe (Pharma-COG partners).
2. Apply the common MRI protocol on phantoms and human subjects to characterize, compare and minimize test-retest variability across the MR sites of WP5 for all the quantitative metrics that will be later assessed on patients.

PART B: By collecting clinical, biochemical, neuroimaging, neuropsychological and neurophysiological data in Mild Cognitive Impairment patient, we aim to:

1. To develop a biomarker MATRIX (made of a combination of biological secondary endpoints) which is more sensitive than the changes observed in the loss of hippocampal volume (primary endpoint) and correlate with the neuropsychological progression and conversion (clinical secondary endpoints).
2. To develop a biomarker MATRIX (made of a combination of biological secondary endpoints) at baseline which is more predictive of the loss of hippocampal volume (primary endpoint) and neuropsychological progression (clinical secondary endpoint) in MCI patients.
3. To harmonize the biomarker MATRIX collection and qualify multiple centres across Europe

ELIGIBILITY:
Inclusion Criteria:

* PART A:

Participants will be (i) healthy volunteers (between 50 and 80 years old) and/or (ii) subjects (between 50 and 80 years old), who will perform a 3T-MRI for reasons such as migraine, headache, auditory or visual symptoms, paresthesias, and whose scan will be negative (see exclusion criteria below). Such subjects will be selected and asked to perform additional sequences according to the part A study protocol.

* PART B:

Specific inclusion criteria:

1. Written Informed Consent to participate in a up to 3 year imaging study
2. Male and female aged between 55-90 years
3. Memory complaint by patient or partner that is verified by a physician. (Memory complains expressed by the patients or their informant that the examiner considers to be relevant and exceed those expected for a patient of their age. The patient may or may not have symptoms of deficiency in other cognitive areas.)
4. Abnormal memory functions documented by scoring 1 SD below the age-adjusted mean on the Logical Memory II subscale, (Delayed Paragraph Recall) from the Wechsler Memory Scale.
5. General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit.
6. Mini-Mental State Exam score between 24 and 30 (inclusive)
7. Clinical Dementia Rating = 0.5. Memory Box score must be at least 0.5.
8. Amnestic Mild Cognitive Impairment (MCI) (pure amnestic or multidomain)
9. Geriatric Depression Scale less than 6
10. Hachinski Modified Ischemic scale< to 4
11. Patient is untreated or under a permitted medication (Cholinesterase inhibitors and memantine, before the enrolment and newly prescriptions during the study, are permitted for aMCI patients.)
12. At least 5 grades education
13. Must speak (language) fluently
14. Have a study partner with 10+ hr/wk contact (can be in person and telephone), accompanies to visits
15. Willing and able to comply with the requirements of the study, as judged by the investigator

Exclusion Criteria:

* PART A:

  1. Ischaemic lesions already detected in a previous scan
  2. Head injury with loss of consciousness > 24 hours
  3. Current substance abuse
  4. Current therapy with steroids or current chemotherapy
  5. Loss of weight > 5 kg in the last 6 months
  6. Systemic disease with frequent involvement of the CNS (lupus, HIV, rheumatoid arthritis)
  7. CNS disease diagnosed by a specialist or in treatment (such as epilepsy, ictus)
  8. Cerebral metastasis or CNS primary tumour still benign (except for pituitary microadenoma)
  9. Suspected multiple sclerosis + MRI evidence of white matter lesions
  10. Suspected recent stroke + MRI evidence of infarct
  11. Aneurysm > 10 mm and arteriovenous malformations (except for venous angioma)
  12. Dysgenesia of central nervous system
* PART B:

  1. Visual and auditory acuity inadequate for neuropsychological testing
  2. Enrolment in other trials or studies not compatible with study objectives (in particular, those with experimental drugs)
  3. History of significant neurological or psychiatric illnesses or presence of other diseases precluding enrolment.
  4. Use of forbidden medications
  5. Ferromagnetic implants and devices not eligible for MRI scanning. Brain malformation or other conditions that may complicate lumbar puncture
  6. Excluded Medication: Antidepressants with anti-cholinergic properties and within 4 weeks of the screening: Regular use of narcotic analgesics (>2 doses per week), Use of neuroleptics with anti-cholinergic properties (e.g., chlorpromazine, thioridazine), Chronic use of other medications with significant central nervous system anticholinergic activity (e.g., diphenhydramine), Use of Anti-Parkinsonian medications (including Sinemet, amantadine, bromocriptine, pergolide, selegiline), Participation in any other investigational drug study (individuals may not participate in any drug study while participating in this protocol). Diuretic drugs should not be started or discontinued within 4 weeks prior to screening (Any change in diuretic medication during the study should be reported).

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2011-12; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Part A: Magnetic Resonance Imagery protocol | Two times: One measure at day 1
  The Magnetic Resonance Imagery protocol comprises a localiser or scout run, 4 structural-volumetric MRI sequences (i.e. 2 MP-RAGE, 1 FLAIR and 1 T2*), a resting state functional MRI acquisition (i.e. rsfMRI), a diffusion tensor scan (i.e. DTI) that will be conducted at the magnetic field strength of 3T and a quantitative assessment of brain perfusion changes with a sequence of Arterial Spin Labelling (i.e. ASL) . The field map will be used for geometric distortion correction of the fMRI data.
  The main parameter of "efficacy" will be the reliability of the acquired MRI data (in terms of their correct acquisition and limited variability).
Part B: Changes of the hippocampal volume | 2 or 3 times: every 18 months during 2 or 3 years (T0, T18 and/or T36)
  The primary endpoint will be changes of the hippocampal volume between the two groups (differentiated by the level of amyloid β1-42 in the cerebro-spinal fluid) and within the same group over time.

SECONDARY OUTCOMES:
Part B: Clinical assessment | Every 6 months (screening, T6, T12, T18, T24, T30 and T36)
  * Mini-Mental State Examination (MMSE) (general cognitive functioning)
  * Clinical Dementia Rating (CDR)
  * Medical History
  * Physical exam
  * Neurological exams
  * Hachinski ischemic scale (differentiate Alzheimer's type dementia and multi-infarct dementia)
  * Geriatric Depression Scale (Depressive symptoms)
  * Functional Assessment Questionnaire (FAQ) (Activities of daily living)
  * Neuropsychiatric Inventory Questionnaire (NPI-Q) (Behaviour)
Part B: Neuropsychology | Every 6 months (screening, T6, T12, T18, T24, T30 and T36)
  * ADAS-COG
  * Clock Drawing and Copying Test (Executive functions and planning abilities)
  * Rey Auditory Verbal Test (AVLT) (Memory)
  * Logical Memory Test I - Immediate Recall (Memory)
  * Digit Span Forward (Memory)
  * Digit Span Backward (Memory)
  * CANTAB Battery (visuospatial functions)
  * Letter fluency (Language)
  * Category Fluency (Language)
  * Boston Naming Test (BNT) (Language)
  * Trail Making Test (Attention)
  * Digit Symbol Substitution Test (Processing speed)
Part B: Neurophysiology | Every 6 months (T0, T6, T12, T18, T24, T30 and T36)
  Electro-Encephalography in several conditions
Part B: Magnetic Resonance Imagery and functional MRI | Every 6 months (screening, T0, T6, T12, T18, T24, T30 and T36)
  The protocol comprises a localiser or scout run, 2 structural-volumetric MRI sequences (i.e. MPRAGE and FLAIR), one 2D structural analysis (i.e. T2*) a resting state functional MRI acquisition (i.e. rs-fMRI), a diffusion tensor scan (i.e. DTI) that will be conducted at the magnetic field strength of 3T and a quantitative assessment of brain perfusion changes with a sequence of Arterial Spin Labelling (i.e. ASL only in T18 and T24 timepoints for available patients).
Part B: Blood drawing | Every 6 months
  * ApoE (T0 only)
  * β amyloid in plasma (T0, T6, T12, T18, T24, T30 and T36)
  * Plasma and lymphocytes biomarkers (T0, T6, T12, T18, T24, T30 and T36)
  * PKC conformation (T0 and T18/T36)
  * amyloid β1-42 binding on erythrocytes (T0 and T18/T36)
  * Platelet APP-CTF (intracellular APP metabolites)(T0, T6, T12, T18, T24, T30 and T36)
  * RNA splicing analysis (T0, T6, T12, T18, T24, T30 and T36)
Part B: Actigraphy | Every 6 months (T0, T6, T12, T18, T24, T30 and T36)
  Assessment of changes in position and acceleration for up to several weeks providing measures of activity. Additionally, sleep/wake and circadian rhythmicity can objectively be estimated from the recorded data by algorithms.
Adverse events | Every 6 months (T0, T6, T12, T18, T24, T30 and T36)
  Any changes in the chronicity, severity, action taken, seriousness of a symptom or adverse event will be recorded by a qualified clinician (MD).

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Frisoni, MD, MP, Study Director — Istituto di Ricovero e Cura a Carattere Scientifico, San Giovanni di Dio Fatebenefratelli, Brescia, Italy; Mira Didic, MD, Principal Investigator — Université de la Méditerranée, Service de Neurologie et Neuropsychologie, Marseille France; Jose-Luis Molinuevo, PhD, Principal Investigator — Institut d'Investigacions Biomèdiques August Pi I Sunyer, Barcelona, Spain; Regis Bordet, MD, Principal Investigator — Université Lille 2, Lille, France; Pierre Payoux, MD, Principal Investigator — Institut National de la Santé et de la Recherche Médicale, Toulouse, France; Peter Schönknecht, MD, Principal Investigator — Universitätsklinikum Leipzig, Department of Psychiatry and Nuclear Medicine, Leipzig, Germany; Jens Wiltfang, MD, Principal Investigator — Universitaet Duisburg-Essen, Department of Psychiatry and Nuclear Medicine, Duisburg-Essen, Germany; Flavio Mariano Nobili, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino-IST; Magda Tsolaki, MD, Principal Investigator — Greek Association of Alzheimer's disease and related disorders, Thessaloniki, Greece; Lucilla Parnetti, MD, Principal Investigator — Università di Perugia, Clinica Neurologica, Centro Disturbi della Memoria, Perugia, Italy; Paolo Maria Rossini, MD, Principal Investigator — Università Cattolica del Sacro Cuore, Policlinico Agostino Gemelli, Istituto di Neurologia, Roma, Italy; Andrea Soricelli, MD, Principal Investigator — Istituto di Ricerca Diagnostica e Nucleare, University of Naples Parthenope, Napoli, Italy; Philip Scheltens, MD, Principal Investigator — VUmc Alzheimercentrum
Locations (13):
- France (3):
  - Université Lille 2, UL2 - Centre d'investigation clinique / Centre de Ressources biologiques 9301 - INSERM - Centre Hospitalier Régional et Universitaire de LILLE, Lille
  - APHM, Hopital de la Timone, Service de Neurologie et Neuropsychologie, Marseille
  - INSERM - CHU Purpan, Toulouse
- Germany (2):
  - Hospital and Institute of the University of Duisburg and Essen - Department for Psychiatry and Psychotherapy, LVR Hospital Essen, Essen
  - University Hospital of Leipzig - Department of Psychiatry, Leipzig
- Aristotle University of Thessaloniki, Greek Association of Alzheimer's disease and related disorders, Thessaloniki, Greece, Thessaloniki, Greece
- Italy (5):
  - IRCCS-FBF - Ordine Ospedaliero San Giovanni di Dio, Fatebenefratelli, Istituto di Ricovero e Cura a Carattere Scientifico, Brescia, Provincia Lombardo-Veneta
  - Neurofisiologia Clinica IRCCS Azienda Ospedaliera Universitaria San Martino-IST, Padiglione Specialita' piano Fondi, Genoa
  - IRCCS Fondazione SDN per la Ricerca e l'Alta Formazione in Diagnostica Nucleare di Napoli, Napoli
  - Dipartimento di Specialità medico-chirurgiche e Sanità Pubblica, Sezione di Clinica Neurologica, Centro Disturbi della Memoria, Perugia, Italy, Perugia
  - Università Cattolica del Sacro Cuore - Policlinico Agostino Gemelli Istituto di Neurologia - Neuropsychological and Neurorehabilitation Unit, Roma
- VUmc Alzheimercentrum, Amsterdam, Netherlands
- Institut d'Investigacions Biomèdiques August Pi I Sunyer, IDIBAPS, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Grady CL, Haxby JV, Horwitz B, Sundaram M, Berg G, Schapiro M, Friedland RP, Rapoport SI. Longitudinal study of the early neuropsychological and cerebral metabolic changes in dementia of the Alzheimer type. J Clin Exp Neuropsychol. 1988 Oct;10(5):576-96. doi: 10.1080/01688638808402796. PMID 3265710
- See also: The Alzheimer-Europe announcement webpage dedicated to PharmaCog project — http://www.alzheimer-europe.org/EN/Research/PharmaCog